CLINICAL TRIAL: NCT04398134
Title: A Phase 2a, Multicenter, Single-Blind, Placebo-Controlled, Multiple Cohort Study Evaluating ABI-H2158-Containing Regimens in Chronic Hepatitis B Infection
Brief Title: A Study of ABI-H2158-containing Regimens in Participants With Chronic Hepatitis B Virus Infection
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to a safety signal of drug-induced liver injury in subjects receiving 2158
Sponsor: Assembly Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABI-H2158-201; 2019-004902-85 (EudraCT Number)
Record Dates: First submitted 2020-05-18; First posted 2020-05-21 (Actual); Results first posted 2022-08-26 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-08

CONDITIONS: Chronic Hepatitis B
Keywords: HBV; hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ABI-H2158 plus ETV (Experimental): ABI-2158 300 mg tablet once daily for 72 weeks plus ETV 0.5 mg tablet once daily for 96 weeks
  Interventions: Drug: ABI-H2158; Drug: Entecavir (ETV)
- Placebo plus ETV (Placebo Comparator): Placebo matching ABI-2158 300 mg tablet once daily for 72 weeks plus ETV 0.5 mg tablet once daily for 96 weeks
  Interventions: Drug: Placebo; Drug: Entecavir (ETV)

INTERVENTIONS:
Drug: ABI-H2158 — 3 X 100 mg tablets for oral administration
  Arms: ABI-H2158 plus ETV
Drug: Placebo — Sugar pill manufactured to mimic the ABI-H2158 tablets
  Arms: Placebo plus ETV
Drug: Entecavir (ETV) — 0.5 mg tablet for oral administration

SUMMARY:
This Phase 2a study will assess the safety, antiviral activity, and pharmacokinetics (PK) of ABI-H2158 administered once daily for up to 72 weeks in combination with entecavir (ETV) in participants with chronic hepatitis B virus (HBV) infection.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18 - 36 kg/m^2 and body weight ≥45 kg
* HBeAg ≥500 IU/mL at Screening
* In good general health except for chronic HBV infection for ≥6 months documented, for example, by at least two measurements of HBsAg positivity and/or detectable HBV DNA ≥6 months apart
* Lack of cirrhosis or advanced liver disease

Exclusion Criteria:

* Prior treatment for chronic HBV infection with lamivudine, telbivudine, adefovir, standard of care nucleoside or nucleotide analogue (NrtI), HBV core inhibitors, or an investigational agent for HBV infection
* History or evidence of advanced liver disease or hepatic decompensation (including jaundice, ascites, portal hypertension, gastrointestinal bleeding, esophageal varices, hepatic encephalopathy)
* History or presence of clinically significant medical conditions requiring frequent medical management or pharmacologic or surgical treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace Wang, Study Director — Assembly Biosciences
Locations (44):
- United States (13):
  - Coalition of Inclusive Medicine, Los Angeles, California
  - California Liver Research Institute, Pasadena, California
  - Stanford University Medical Center, Redwood City, California
  - Research and Education Inc., San Diego, California
  - Quest Clinical Research, San Francisco, California
  - University of Miami/Schiff Center for Liver Diseases, Miami, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - New Discovery, LLC, Flushing, New York
  - Northwell Health Center for Liver Disease, Manhasset, New York
  - NYU Langone Health, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
  - University of Washington, Seattle, Washington
- Australia (7):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Gallipoli Medical Research Foundation, Greenslopes, Queensland
  - St. Vincent's Hospital, Fitzroy, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Melbourne Health, Parkville, Victoria
- Canada (2):
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Toronto Liver Centre, Toronto, Ontario
- China (5):
  - The First Hospital of Jilin University, Changchun, Jilin
  - The Second Affliated Hospital of Chongqing Medical University, Chongqing, Yuzhong District
  - Xiangya Hospital Central South University, Changsha
  - Nanfang Hospital, Guangzhou
  - Guangzhou Eighth People's Hospital - Guangzhou Infectious Diseases Hospital, Guangzhou
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - Queen Mary Hospital, Hong Kong
- New Zealand (2):
  - Auckland Clinical Studies, Auckland
  - Waikato Hospital, Hamilton
- South Korea (7):
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Kaohsiung City, Sanmin District
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital Taipei Branch, Taipei
  - Chang Gung Memorial Hospital (CGMH) - Linkou Branch, Taoyuan District
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ABI-H2158 Plus ETV (HBeAg Positive Population); ABI-H2158 Plus ETV (HBeAg Negative Population): ABI-2158 300 mg tablet once daily for 72 weeks plus ETV 0.5 mg tablet once daily for 96 weeks
  ABI-H2158: 3 X 100 mg tablets for oral administration
  Entecavir (ETV): 0.5 mg tablet for oral administration
- Placebo Plus ETV (HBeAg Positive Population); Placebo Plus ETV (HBeAg Negative Population): Placebo matching ABI-2158 300 mg tablet once daily for 72 weeks plus ETV 0.5 mg tablet once daily for 96 weeks
  Placebo: Sugar pill manufactured to mimic the ABI-H2158 tablets
  Entecavir (ETV): 0.5 mg tablet for oral administration
Period: Overall Study
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Started | 32 | 11 | 33 | 12
Completed | 0 | 0 | 0 | 0
Not Completed | 32 | 11 | 33 | 12
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1
Not completed — Study Terminated by Sponsor | 30 | 11 | 32 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population) | Total
Number analyzed (Participants) | 32 | 11 | 33 | 12 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (8.3) | 35 (9.8) | 44 (11) | 46 (9.8) | 41 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 13 | 8 | 40
  Male | 19 | 5 | 20 | 4 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 32 | 10 | 31 | 12 | 85
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 2
  White | 0 | 1 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  New Zealand | 1 | 1 | 1 | 0 | 3
  Canada | 0 | 0 | 3 | 1 | 4
  South Korea | 4 | 0 | 3 | 0 | 7
  Hong Kong | 8 | 3 | 5 | 3 | 19
  United States | 8 | 2 | 8 | 3 | 21
  China | 6 | 2 | 10 | 4 | 22
  Taiwan | 4 | 1 | 3 | 1 | 9
  United Kingdom | 1 | 2 | 0 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events
Description: Describes the number of participants with One or More Adverse Events while they were on treatment with the study drug.
Time Frame: Up to 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 32 | 11 | 33 | 12
Participants | 18 | 6 | 19 | 6

2. Primary Outcome: Percentage of Participants With Premature Treatment Discontinuation
Description: Describes the number of participants who discontinued treatment with ABI-H2158/placebo prematurely.
Time Frame: Up to 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 32 | 11 | 33 | 12
Participants | 2 | 0 | 2 | 0

3. Primary Outcome: Change From Baseline in Mean log10 HBV DNA
Description: HBV DNA was measured by Cobas AmpliPrep/ Cobas TaqMan HBV Test v2.0 (LOD 10 IU/mL). The analysis of data was descriptive only.
Time Frame: Baseline and Week 24
Population: Due to early termination of the study, samples at Week 24 from participants in the HBeAg negative cohort were not collected.
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 5 | 2 | 0 | 0
log10 IU/mL | -6.2 (0.76) | -4.8 (0.25) |  |

4. Primary Outcome: Percentage of Participants With Abnormal Laboratory Results
Description: Severity grades were defined by Grading Scale for Severity of Adverse Events and Laboratory Abnormalities [The DAIDS Version 2.1]. For maximum postbaseline toxicity grade, the most severe graded abnormality from all tests was counted for each participant. For each individual laboratory test, the most severe graded abnormality for that test was counted for a participant. A treatment-emergent laboratory abnormality was defined as an increase of at least 1 toxicity grade from baseline at any time postbaseline up to and including the date of last dose of ABI-H2158/Placebo plus 28 days.
Time Frame: Up to 72 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 32 | 11 | 33 | 12
Participants | 29 | 8 | 19 | 9

5. Secondary Outcome: Trough Plasma Concentration of ABI-H2158
Time Frame: Predose on Day 1, Week 4, Week 48, and Week 72
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: Trough-to-Peak Plasma Concentration Ratio of ABI-H2158
Time Frame: Predose on Day 1 and Weeks 4, 48, and 72 and at pre-specified intervals after dosing on Day 1 and Weeks 2, 8, 12, 16, 20, 24, and 28
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Trough Plasma Concentration of ETV
Time Frame: Predose on Day 1, Week 4, Week 48, and Week 72
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Trough-to-Peak Plasma Concentration Ratio of ETV
Time Frame: as for outcome 6
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Change in Mean log10 HBV pgRNA From Baseline to Week 24 and at Each Timepoint for ABI-H2158+ETV and PBO+ETV
Time Frame: up to Week 72
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Reduction in HBV DNA Below the Assay Lower Limit of Quantitation
Time Frame: Up to 72 weeks
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Reduction in HBV pgRNA Below the Assay Lower Limit of Quantitation
Time Frame: Up to 72 weeks
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

12. Secondary Outcome: Change From Baseline in Serum HBV Surface Antigen (HBsAg)
Time Frame: Baseline and up to 72 weeks
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Change From Baseline in Serum HBV "e" Antigen (HBeAg)
Time Frame: Baseline and up to 72 weeks
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Change From Baseline in Serum HBV Core-related Antigen (HBcrAg)
Time Frame: Baseline and up to 72 weeks
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Proportion of Subjects With Abnormal ALT at Baseline Who Have Normal ALT at Week 24 and at Each Timepoint on ABI-H2158+ETV and PBO+ETV
Time Frame: Baseline and up to Week 24
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Ncidence of HBV Variants With Reduced Susceptibility to ABI-H2158
Time Frame: Up to 72 weeks
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Change in Mean log10 HBV DNA for ABI-H2158+ETV and PBO+ETV at Each Timepoint
Time Frame: up to 72 weeks
Population: Due to early termination of the study, data were not collected and analyzed for secondary outcomes.
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 72 weeks
Arm/Group | ABI-H2158 Plus ETV (HBeAg Positive Population) | Placebo Plus ETV (HBeAg Positive Population) | ABI-H2158 Plus ETV (HBeAg Negative Population) | Placebo Plus ETV (HBeAg Negative Population)
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/11 | 0/33 | 0/12
Serious Adverse Events (participants affected / at risk) | 1/32 | 1/11 | 0/33 | 1/12
Other Adverse Events (participants affected / at risk) | 18/32 | 6/11 | 19/33 | 6/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABI-H2158 Plus ETV (HBeAg Positive Population) (N=32) | Placebo Plus ETV (HBeAg Positive Population) (N=11) | ABI-H2158 Plus ETV (HBeAg Negative Population) (N=33) | Placebo Plus ETV (HBeAg Negative Population) (N=12)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ABI-H2158 Plus ETV (HBeAg Positive Population) (N=32) | Placebo Plus ETV (HBeAg Positive Population) (N=11) | ABI-H2158 Plus ETV (HBeAg Negative Population) (N=33) | Placebo Plus ETV (HBeAg Negative Population) (N=12)
alanine aminotransferase increased (Investigations) | 5 | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 2 | 0
headache (Nervous system disorders) | 1 | 1 | 3 | 1
diarrhea (Gastrointestinal disorders) | 0 | 0 | 3 | 1
abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 0
white blood cell count decreased (Investigations) | 0 | 0 | 2 | 0
hyperuricaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2
hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
vaccination complication (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1
folliculitis (Infections and infestations) | 0 | 1 | 0 | 0
anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Hyperlactacidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
International Normalised Ratio Increased (Investigations) | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Libido Increased (Psychiatric disorders) | 0 | 1 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 1
Malaise (General disorders) | 1 | 0 | 0 | 0
Menstruation Delayed (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Mesenteric Panniculitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Monocyte Count Increased (Investigations) | 0 | 0 | 1 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 1 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 1 | 0
Poor Quality Sleep (Nervous system disorders) | 1 | 0 | 0 | 0
Post Vaccination Syndrome (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Prothrombin Time Prolonged (Investigations) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Supraventricular Extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tibia Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Viral Infection (Infections and infestations) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1
Chest Pain (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0 | 1 | 0
Amylase Increased (Investigations) | 0 | 0 | 0 | 1
Blood Bilirubin Increased (Investigations) | 1 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 1 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Altered State Of Consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Study ABI-H2158-201 was terminated early due to alanine aminotransferase (ALT) elevations among study participants who received ABI-H2158 (and not among those who received PBO). Further details on these events are described in the results section below. In the absence of an alternative etiology for the ALT elevations, further clinical development of ABI-H2158 was terminated by the Sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Assembly Biosciences agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Assembly Biosciences supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT04398134/Prot_SAP_000.pdf